CLINICAL TRIAL: NCT02011750
Title: Pilot Trial of Valproate as Adjunctive Treatment for Toxoplasma Gondii
Brief Title: Pilot Trial of Valproate as Adjunctive Treatment for Toxoplasma Gondii Infection in Early Course Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Mansoura University (Other); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Hader Mansour, MD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO12020320
Record Dates: First submitted 2013-06-21; First posted 2013-12-13 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Toxoplasmosis; Schizophrenia
Keywords: schizophrenia; toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis; Schizophrenia | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Valproate treatment (Experimental): Sodium Valproate treatment:During the entry period, all patients will have a placebo run-in for two weeks after which they will be evaluated for the outcome variables and then randomized to either Sodium Valproate (Depakote, DEP) or placebo (PLA) group in a 1:1 proportion. For the Sodium Valproate treatment grou, this will be followed by a two week period to adjust the dose of DEP and attain therapeutic levels (50-100 µg/mL). Then DEP treatment will continue for 16 more weeks, after which DEP will be discontinued. Subject will be followed up for four weeks post-DEP discontinuation to monitor delayed adverse side effects.
  Interventions: Drug: Sodium Valproate treatment; Drug: Placebo
- Placebo (Placebo Comparator): Placebo Comparator: During the entry period, all patients will have a placebo run-in for two weeks after which they will be evaluated for the outcome variables and then randomized to either the experimental Sodium Valproate (Depakote, or DEP) or placebo (PLA) group in a 1:1 proportion. For the PLA group, this will be followed by a two week period of placebo during which members of the experimental Sodium Valproate (Depakote/DEP) will have DEP dose adjusted to attain therapeutic levels (50-100 µg/mL). Then PLA treatment will continue for 16 more weeks. Subjects will be followed up for four weeks post PLA-discontinuation to monitor for delayed adverse side effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Valproate treatment — Sodium Valproate treatment:During the entry period, all patients will have a placebo run-in for two weeks after which they will be evaluated for the outcome variables and then randomized to either Sodium Valproate (Depakote, DEP) or placebo (PLA) group in a 1:1 proportion. For the Sodium Valproate treatment group, this will be followed by a two week period to adjust the dose of DEP and attain therapeutic levels (50-100 µg/mL). Then DEP treatment will continue for 16 more weeks, after which DEP will be discontinued. Subject will be followed up for four weeks post-DEP discontinuation to monitor delayed adverse side effects.
  Other Names: Depakote
  Arms: Sodium Valproate treatment
Drug: Placebo — Placebo: During the entry period, all patients will have a placebo run-in for two weeks after which they will be evaluated for the outcome variables and then randomized to either the experimental Sodium Valproate (Depakote, or DEP) or placebo (PLA) group in a 1:1 proportion. For the PLA group, this will be followed by a two week period of placebo during which members of the experimental Sodium Valproate (Depakote/DEP) will have DEP dose adjusted to attain therapeutic levels (50-100 µg/mL). Then PLA treatment will continue for 16 more weeks. Subjects will be followed up for four weeks post PLA-discontinuation to monitor for delayed adverse side effects.

SUMMARY:
This is an exploratory study in Egypt that will combine a treatment trial among early course schizophrenia (ECSZ) patients with key analyses suggested by rodent studies. Specifically, the study will test the provocative results from animal studies indicating an impact of Toxoplasma Gondii (TOX) exposure on novelty seeking. The study will also test whether exposure to TOX is associated with other cognitive and behavioral changes, as well as changes in overall social function. We will also explore the relative efficacy of Sodium Valproate (Depakote, DEP) in improving clinical and overall social function among TOX exposed and unexposed patients.

Hypotheses

1. At baseline, TOX exposure is associated with increased novelty seeking, clinical severity, and impaired cognitive and overall social function in patients with SZ.
2. Adjunctive DEP treatment improves clinical symptoms, cognitive and social function in SZ, particularly among TOX exposed SZ patients.
3. Exploratory hypothesis: adjunctive DEP reduces serological indices of TOX infection (VIP and TH levels).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult men or women (ages 18-50 years)
* Schizophrenia / schizoaffective disorder (DSM IV)
* Duration of illness < 5 years (since onset of psychosis)
* On a stable dose of an antipsychotic for at least a month
* Scores 4 or more on at least one item of the Positive and Negative Syndrome Scale.

Exclusion Criteria:

* Substance abuse in the past month/dependence past 6 months
* History of / or current medical/neurological illnesses e.g. mental retardation (DSM-IV) or epilepsy;
* Medical conditions that are judged by the consulting internist and research staff to be unstable
* Pregnant or breast-feeding women
* Known allergy or serious adverse event to DEP, Received Chlorpromazine, Trimethoprim or DEP for up to 6 months prior to study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Severity | Clinical severity will be assessed during week 20 of the study.
  Clinical Severity will be measured by the Positive and Negative Syndrome Scale (PANSS),a 7 point rating scale for 30 psychopathological items based on interviews or reports.
Cognitive Domains assessed via the Arabic version of the Penn CNB | Cognitive domains wil be measured in week 16 of the study
  Cognitive domains will be assessed using the Arabic version of the Penn Computerized Neuropsychological Battery (CNB), which includes cognitive measures that distinguish SZ cases and relatives from controls. Accuracy and response time are recorded.
Social Function assessed via the Quality of Life Scale | Social functioing will be assessed during week during week 16.
  Overall Social function will be measured by the Quality of Life Scale, which measures interpersonal, social and occupational functioning.
Cognitive domains assessed via Trails Making Test | Cognitive domains will be assessed in week 16 of the study
  Cognitive domains will be assessed using the Trails Making Test, a neuropsychological test of attention and task switching.
Social Function -assessed via the GAF scale | Social functioning will be assessed during week 16
  Social functioning will be assessed using the Global Assessment of Functioning (GAF), a global measure of function and symptom severity.
Social Functioning assessed via the Short Form | Social functioning will be assessed during week 16
  Social functioning will be assessed via the Short Form, a multi-item scale that consists of 8 scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.

SECONDARY OUTCOMES:
Side effects | Side effects will be measured during week 20 of the study.
  Participants will be monitored for adverse reactions to study medication through week 20.

CONTACTS AND LOCATIONS:
Overall Officials: Hader Mansour, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt